CLINICAL TRIAL: NCT02888119
Title: Imaging Biomarkers of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-00918
Record Dates: First submitted 2016-08-26; First posted 2016-09-02 (Estimated); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- High Risk for Osteoarthritis (Active Comparator): "High risk of developing knee OA" has been defined by having knee pain but normal radiographs (Kellgren-Lawrence score 0 i.e. KL0) on both knees but at least one abnormal finding on clinical MR protocol such as overweight, prior knee injury (ligaments or menisci) or traumatic bone marrow edema lesions.
  Interventions: Device: PRISMA 3T MRI scanner (Siemens Medical Solutions)
- Mild Osteoarthritis (Active Comparator)
  Interventions: Device: PRISMA 3T MRI scanner (Siemens Medical Solutions)
- Healthy Controls (Active Comparator): Controls will be age/gender matched to patients within 2 years of age.
  Interventions: Device: PRISMA 3T MRI scanner (Siemens Medical Solutions)

INTERVENTIONS:
Device: PRISMA 3T MRI scanner (Siemens Medical Solutions) — A baseline MRI exam consisting of accelerated 3D-T1p, and T2, MRI will be performed. Longitudinal follow-up MRI exams (24 months) will be repeated on the same knee on all OA patients.

SUMMARY:
This study aims to develop, evaluate and translate highly accelerated imaging sequences (each protocol under 5 minutes) for in-vivo knee Osteoarthritis applications on a standard clinical 3T scanner using novel compression sensing and parallel imaging strategies.The overarching objective of the study is to establish a non-invasive imaging biomarker based on the development of rapid relaxation mapping with compressed sensing (CS) that will be clinically useful for assessment of early Osteoarthritis. A total of 90 subjects including 30 patients with high risk of developing knee osteoarthritis (OA), 30 patients with mild OA and 30 healthy controls will be accrued.

DETAILED DESCRIPTION:
Current noninvasive imaging methods to evaluate knee joints include plain radiographs, computed tomography (CT), and clinical morphological magnetic resonance imaging (MRI) of joint structures. These techniques can only detect later-stage, macroscopic joint structural abnormalities that are irreversible and not amenable to early therapy. This study aims to develop highly accelerated imaging sequences for ex-vivo knee OA applications on a standard clinical 3T scanner using novel CS and parallel imaging (PI) strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the HJD OA database, ages 40-75 with high risk of developing OA as defined by:

  (i) KL score of 0 (ii) Knee pain present in at least 1 knee (iii) Normal radiographs, (iv) At least one abnormal clinical MR finding such as prior knee injury, overweight or traumatic bone marrow edema lesions
* Patients ages 40-75 with early OA as determined by KL scores 1-2
* Healthy controls in the HJD OA database (KL score 0, no knee pain, no meniscal or ligament tears)

Exclusion Criteria:

* Contraindications for MRIs (e.g. pacemakers, ferromagnetic vascular clips, metal implants, claustrophobia, etc).
* Subjects with any joint disease (example: Rheumatoid or inflammatory arthritis) other than knee OA, corticosteroid injections within the previous 3 months, and history of avascular necrosis, Paget's disease of bone, Wilson's disease, gout, total knee replacement (or plan for replacement within next 24 months).
* Major co-morbidities such as diabetes, mellitus, cancer, congestive heart failure and chronic infectious diseases.
* Alignment interventions such as insoles and knee braces
* Vulnerable patients will not be recruited for this study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Regatte, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Controls will be age/gender matched to patients within 2 years of age.
  PRISMA 3T MRI scanner (Siemens Medical Solutions): A baseline MRI exam consisting of accelerated 3D-T1p, and T2, MRI will be performed.
Period: Overall Study
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis | Healthy Controls
Started | 11 | 7 | 30
Completed | 6 | 3 | 30
Not Completed | 5 | 4 | 0
Not completed — Lost to Follow-up | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis | Healthy Controls | Total
Number analyzed (Participants) | 6 | 3 | 30 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (4.5) | 64.7 (5.7) | 57.9 (8.6) | 59.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 15 | 21
  Male | 2 | 1 | 15 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 4 | 2 | 20 | 26
  Unknown or Not Reported | 0 | 1 | 8 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 11 | 12
  White | 4 | 1 | 11 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 30 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in T1ρ Relaxation Time
Description: MRI exam of accelerated 3D-T1p conducted on whole knee joint specimens to determine cartilage composition, measured as T1ρ relaxation time. T1ρ MRI relaxation times refer to the proteoglycan density within cartilage.
  Images taken at baseline and at Month 24.
Time Frame: Baseline, Month 24
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis
Number analyzed (Participants) | 6 | 3
milliseconds | 2.1 (2.2) | 13.3 (9.4)

2. Primary Outcome: Change From Baseline in T2 Relaxation Time
Description: MRI exam of accelerated T2 conducted on whole knee joint specimens to determine cartilage composition, measured as T2 relaxation time. T2 relaxation represents the time constant of the molecular motion of water in cartilage, which is influenced by the composition of collagen and specifically reflects changes to the extracellular matrix. Images taken at baseline and at Month 24.
Time Frame: Baseline, Month 24
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis
Number analyzed (Participants) | 6 | 3
milliseconds | 0.7 (6.3) | 11 (7.8)

3. Secondary Outcome: Change From Baseline in Western Ontario and McMaster University OA Index (WOMAC) Score
Description: The WOMAC is a 33-item self assessment of how participants feel about their knee and how well they can perform usual activities. The questionnaire contains 4 separately scored subscales - Symptoms; Stiffness; Pain and Function; and Daily Living. The total score is a percentage score from 0 to 100; lower scores represent less pain, less stiffness, and better physical function; higher scores indicate greater pain, greater stiffness, and worse physical function. A decrease in scores indicates participants' health improved during the observational period.
Time Frame: Baseline, Month 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis
Number analyzed (Participants) | 6 | 3
score on a scale | 5.4 (8.6) | 2.5 (4.1)

4. Secondary Outcome: Change From Baseline in Knee Injury and OA Outcomes Score (KOOS)
Description: Knee-specific instrument, developed to assess patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales - Pain; Other Symptoms; Function in daily living (ADL); Function in Sport and Recreation (Sport/Rec); and knee-related Quality of Life (QOL). The total score is a percentage score from 0 to 100; 0 represents extreme problems and 100 represents no problems. An increase in scores indicates participants' health improved during the observational period.
Time Frame: Baseline, Month 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis
Number analyzed (Participants) | 6 | 3
score on a scale | 6 (11.9) | 6.2 (4.5)

5. Secondary Outcome: Change From Baseline in Physical Activity Scale for the Elderly (PASE) Scores
Description: Self-assessment of multiple domains of activity in older adults. Questions evaluate both occupational and non-occupational knee bending, squatting and stair climbing. Total scores range from 0 to 400 or above and are quantified based on frequency values and weights for these activities. Higher scores indicate higher levels of physical activity. An increase in scores indicates physical activity increased during the observational period.
Time Frame: Baseline, 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis
Number analyzed (Participants) | 6 | 3
score on a scale | 3.8 (10.1) | 3.2 (4.5)

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | High Risk for Osteoarthritis | Mild Osteoarthritis | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/30
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT02888119/Prot_SAP_000.pdf